CLINICAL TRIAL: NCT04993703
Title: Comparison of Short-term Effect of the Kinesiotaping and Night Splinting in Patients With Carpal Tunnel Syndrome
Brief Title: Effect of Kinesiotaping and Night Splinting in Patients With Carpal Tunnel Syndome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Leyla Eraslan, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HEK 12/57
Record Dates: First submitted 2021-07-08; First posted 2021-08-06 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; night splinting; kinesiotaping; physiotherapy and rehabilitation
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesiotaping (Experimental): A total of 20 sessions physiotherapy sessions including hot pack, ultrasound and exercise program (tendon and nerve gliding exercises=2 times per day 3sets of ten repetitions) will be applied.
  Additionally for this group, kinesiotaping will be applied by using carpal tunnel technique including button hole and I band technique of space correction; and with 25-50% tension in center of tape over dorsal carpal tunnel at the end of the each session. Patients will request to keep kinesiotaping at nights throughout the study.
  Interventions: Other: Kinesiotaping
- Night splinting (Experimental): A total of 20 sessions physiotherapy sessions including hot pack, ultrasound and exercise program (tendon and nerve gliding exercises=2 times per day 3sets of ten repetitions) will be applied.
  Additionally, night splinting will be advised. Patients will request to keep their splints at nights throughout the study.
  Interventions: Other: Night Splinting
- Control group (Experimental): A total of 20 sessions physiotherapy sessions including hot pack, ultrasound and exercise program (tendon and nerve gliding exercises=2 times per day 3sets of ten repetitions) will be applied.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Kinesiotaping — A total of 20 sessions physiotherapy sessions including hot pack, ultrasound, kinesiotaping and exercise program (tendon and nerve gliding exercises=2 times per day 3 sets of ten repetitions) will be applied.times per day 3sets of ten repetitions) will be applied.
  Arms: Kinesiotaping
Other: Night Splinting — A total of 20 sessions physiotherapy sessions including hot pack, ultrasound, night splinting and exercise program (tendon and nerve gliding exercises=2 times per day 3 sets of ten repetitions) will be applied.
  Arms: Night splinting
Other: Control Group — A total of 20 sessions physiotherapy sessions including hot pack, ultrasound and exercise program (tendon and nerve gliding exercises=2 times per day 3 sets of ten repetitions) will be applied.
  Arms: Control group

SUMMARY:
Carpal tunnel syndrome (CTS) which is defined as a symptomatic compression neuropathy of the median nerve at the level of the wrist.

Different types of splints are used for improving the function and decreasing the pain intensity and symptoms in the rehabilitation of patients with CTS.

However effectiveness of treatment by taping has never been investigated in physiotherapy and rehabilitation.

The aim of this study was to compare the short-term effect of conventional physiotherapy only, and also kinesio taping and night splinting in patients with CTS.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) which is defined as a symptomatic compression neuropathy of the median nerve at the level of the wrist.It is considered as the most common disabling neuromuscular condition of the upper extremities.

Night splints are used in conjunction with the conservative intervention to improve the function and decrease the pain intensity and paresthesia in the rehabilitation of patients with carpal tunnel syndrome. However effectiveness of treatment by kinesiotaping has never been investigated.

The aim of this study was to compare the short-term effect of conventional physiotherapy only, and also kinesio taping and night splinting in addition to conventional physiotherapy in the rehabilitation of patients with CTS.

ELIGIBILITY:
Inclusion Criteria:

* This study included patients with moderate CTS, confirmed by electroneurographic examination.
* did not recruit any treatment (including physiotherapy or surgical release)

Exclusion Criteria:

* Patients suffer from the thenar muscle atrophy.
* Patients with mild CTS.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
functional impairment | functional impairment will be recorded at baseline and 4-week follow-up
  functional impairment will be assessed by using Boston Carpal Tunnel Questionnaire. The score consisted of two sub-scales; The Symptom Severity Scale including 11 questions and The Functional Capacity Scale including 8 questions. Each scale score is calculated by the average values of the questions. The scores vary between "1-point" to "5-point". High score indicates severe symptoms and impaired functional capacity.

SECONDARY OUTCOMES:
pain intensity | change from baseline to 4-week follow-up will be recorded
  pain intensity will be assessed by using Visual Analog Scale at rest, activity and at night.
  All patients were asked to mark their pain level that corresponds to their pain intensity on the line between "0=no pain" and "100=the worst pain imaginable".
paresthesia | change from baseline to 4-week follow-up will be recorded
  Paresthesia will be assessed by using Visual Analog Scale at rest, activity and at night.
  All patients were asked to mark their paresthesia level that corresponds to their paresthesia intensity on the line between "0=no paresthesia" and "100=the worst paresthesia imaginable".

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Eraslan L, Baltaci G. Effectiveness of Kinesio Taping and Night Splinting Along With Physical Therapy Intervention on Symptoms and Functionality: A Double-Blind Randomized Controlled Trial for Moderate Carpal Tunnel Syndrome. Am J Phys Med Rehabil. 2023 Nov 1;102(11):975-983. doi: 10.1097/PHM.0000000000002252. Epub 2023 Mar 29. PMID 37026822